CLINICAL TRIAL: NCT04612764
Title: Noninvasive Biomarkers of Hepatic Fibrosis in Urea Cycle Disorders
Brief Title: Liver Disease in Urea Cycle Disorders
Status: Recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: Children's National Research Institute (Other); Seattle Children's Hospital (Other); Children's Hospital Colorado (Other); Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Lindsay Burrage, Principal Investigator, Baylor College of Medicine
Other Study IDs: H-50295
Record Dates: First submitted 2020-10-22; First posted 2020-11-03 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Urea Cycle Disorder; Ornithine Transcarbamylase Deficiency; Citrullinemia 1; ARGI Deficiency; ASL Deficiency; Argininosuccinic Aciduria; ASS Deficiency; Hyperargininemia
Keywords: Liver disease; Fibroscan; Magnetic resonance elastography; Fibrotest
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Ornithine Carbamoyltransferase Deficiency Disease; Citrullinemia; Hyperargininemia; Argininosuccinic Aciduria; Liver Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a multi-center, cross-sectional study to assess risk for liver fibrosis and hepatic injury in individuals with urea cycle disorders (UCDs) using serum biomarkers, Fibroscan, and MRE. This study will be conducted at 5 sites of the Urea Cycle Disorders Consortium: Baylor College of Medicine in Houston, TX, Seattle Children's Hospital in Seattle, WA, Children's Hospital Colorado in Aurora, CO, Children's Hospital of Philadelphia in Philadelphia, PA, and Children's National Medical Center in Washington D.C.

DETAILED DESCRIPTION:
Urea cycle disorders (UCDs) are among the most common inborn errors of liver metabolism. With early diagnosis and improved treatments, the survival of individuals with UCDs has improved, and this improved survival has led to unmasking of some long-term complications such as hepatic dysfunction and progressive fibrosis in a subset of patients. Hepatic complications in UCDs are quite variable and dependent upon the specific metabolic defect.

Currently, there are no guidelines for monitoring hepatic complications or extent of liver disease in UCDs. The gold standard for staging of fibrosis or confirming cirrhosis has traditionally been liver biopsy, an invasive procedure with inherent risks, particularly in the setting of a UCD and compromised coagulation. Recently, non-invasive serum and imaging-based biomarkers have been introduced to assess hepatic fibrosis in adults and children who are at increased risk. Utilization of these technique in individuals with UCDs could be invaluable in both the research and clinical arenas.

The purpose of this study is:

1) To assess risk for increased fibrosis using serum biomarkers and/or VCTE in distal disorders (ASS1D, ASLD and ARG1D) as compared to OTCD 2 ) To assess risk for hepatic fibrosis (liver stiffness as measured by MRE) in individuals with UCDs who have abnormal serum biomarkers and/or VCTE as those who have normal values

ELIGIBILITY:
Stage A

Inclusion Criteria:

* Age > 6 years and < 65 years
* Weight ≥ 11 kg at time of screening
* A molecular or biochemical diagnosis of OTCD, ASS1D, ASLD, or ARG1D.

Exclusion Criteria:

* Prior liver transplantation
* Episode of acute hyperammonemia (≥100 umol/L) in the 30 days prior to enrollment
* Confirmed diagnosis of chronic viral hepatitis, autoimmune liver disease, short gut, small bowel syndrome, alcohol liver disease, TPN requirement, or TPN-related cholestatic disease
* Adults with BMI ≥ 45 kg/m2
* Current pregnancy
* Open wound near expected Fibroscan® probe application site
* Use of implantable active medical device such as cardiac pacemaker or implantable cardioverter-defibrillator

Stage B Inclusion Criteria

• Participation in Stage A of this study

Exclusion Criteria

* Individuals with claustrophobia or other inability to complete
* Known diagnosis of hemochromatosis
* Presence of implants or devices incompatible with MRI
* Inability to breath-hold for 20 seconds for the elastography sequence
* Current pregnancy
* Confirmed diagnosis of chronic viral hepatitis, autoimmune liver disease, short gut, small bowel syndrome, alcohol liver disease, TPN requirement, or TPN-related cholestatic disease
* Episode of documented acute hyperammonemia (ammonia ≥ 100 umol/L) in the 30 days prior to scheduled visit for Stage B

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with urea cycle disorders
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Fibrotest | One measurement made on the 1 day of the study visit (stage A)
  Fibrotest(TM)
Fibroscan (liver stiffness) | One measurement made on the 1 day of the study visit (stage A)
  Liver stiffness (kPa) as assessed by Fibroscan®
Fibroscan (CAP) | One measurement made on the 1 day of the study visit (stage A)
  Controlled Attenuation Parameter (CAPTM in dB/m) as assessed by Fibroscan®
MRE | One measurement made on the 1 day of the study visit (stage B)
  Liver stiffness (kPa) as measured by MRE

SECONDARY OUTCOMES:
Albumin | One measurement made on the 1 day of the study visit (stage A)
  Albumin
Liver Enzymes | One measurement made on the 1 day of the study visit (Stage A)
  Aspartate aminotransferase, Alanine aminotransaminase, and Gamma glutamyl transferase
Total Bilirubin | One measurement made on the 1 day of the study visit (stage A)
  Total Bilirubin
Prothrombin time | One measurement made on the 1 day of the study visit (stage A)
  Prothrombin time
INR | One measurement made on the 1 day of the study visit (stage A)
  INR
AST-to-Platelet Ratio (APRI) | One measurement made on the 1 day of the study visit (stage A)
  AST-to-Platelet Ratio (APRI)
GGT-to-Platelet Ratio (GPR) | One measurement made on the 1 day of the study visit (stage A)
  GGT-to-Platelet Ratio (GPR)
Fibrosis-4 (FIB-4) Index | One measurement made on the 1 day of the study visit (stage A)
  Fibrosis-4 (FIB-4) Index
MRE | One measurement made on the 1 day of the study visit (stage B)
  Fat fraction (%) as measured by MRE

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Burrage, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (5):
- United States (5):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No